CLINICAL TRIAL: NCT01297582
Title: A Double-Blind, Placebo-Controlled, Single-Dose Escalation and Food Effect Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ONO-6950 in Healthy Adult Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ONO-6950 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-6950POU001
Record Dates: First submitted 2011-02-11; First posted 2011-02-17 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Adult Subjects
Keywords: ONO-6950; Healthy Adult Subjects
MeSH Terms: interventions — gemilukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- E (Experimental)
  Interventions: Drug: ONO-6950
- P (Placebo Comparator)
  Interventions: Drug: ONO-6950

INTERVENTIONS:
Drug: ONO-6950 — 1mg, 3mg, 10mg, 30mg,100mg,300mg,1000mg at a single dose; 30mg, 100mg and 300mg for food effect study
  Arms: E
Drug: ONO-6950 — 1mg, 3mg, 10mg, 30mg, 100mg, 300mg, 1000mg at a single dose; 30mg, 100mg and 300mg for food effect study
  Arms: P

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of ONO-6950 across ascending single doses in healthy adult male and female subjects. The secondary objectives are to characterize the pharmacokinetic and pharmacodynamic profiles of ONO-6950 by measuring plasma concentrations of ONO-6950, pulmonary function, and potential cardiovascular effects. The tertiary objective of this study is to evaluate the effect of a meal upon the pharmacokinetic profile of ONO-6950.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male or female subjects (18-55 inclusive)
* Body mass index (BMI) of 19-35kg/m2 (inclusive)
* For females, postmenopausal, non-lactating, and non-pregnant

Exclusion Criteria:

* History or presence of clinical significant disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ONO-6950 using vital signs, pulmonary function tests, ECGs, laboratory tests, physical examinations | up to 7 days

SECONDARY OUTCOMES:
Characterization of PK and PD profiles of ONO-6950, including change from baseline in pulmonary function tests, and any potential cardiovascular effects | up to 7 days
Effect of food on ONO-6950 pharmacokinetics by comparison of PK profile between fasted and fed conditions | up to 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Miramar Clinical Site, Miramar, Florida, United States